CLINICAL TRIAL: NCT02387554
Title: A Randomized, Open-label, 4-way Crossover Single Dose Clinical Trial to Investigate the Pharmacokinetic Interaction Between HGP0904, HGP0608 and HGP1405 When Administered Alone and in Combination in Healthy Male Volunteers
Brief Title: Pharmacokinetic Interaction Between HGP0904, HGP0608 and HGP1405
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HM-ALCH-101
Record Dates: First submitted 2014-12-17; First posted 2015-03-13 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-05

CONDITIONS: Hypertension(HTN)
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Losartan; Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HGP0904+HGP0608+HGP1405 (Experimental): amlodipine + losartan + chlorthalidone
  Interventions: Drug: HGP0904; Drug: HGP0608; Drug: HGP1405
- HGP0904 (Active Comparator): amlodipine
  Interventions: Drug: HGP0904
- HGP0608 (Active Comparator): losartan
  Interventions: Drug: HGP0608
- HGP1405 (Active Comparator): chlorthalidone
  Interventions: Drug: HGP1405

INTERVENTIONS:
Drug: HGP0904
  Other Names: amlodipine
  Arms: HGP0904; HGP0904+HGP0608+HGP1405
Drug: HGP0608
  Other Names: losartan
  Arms: HGP0608; HGP0904+HGP0608+HGP1405
Drug: HGP1405
  Other Names: chlorthalidone
  Arms: HGP0904+HGP0608+HGP1405; HGP1405

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic interaction and safety between HGP0904, HGP0608 and HGP1405 when administered alone and in combination in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* 19~45 years old
* Healthy men

Exclusion Criteria:

* Gastroentestinal disease affecting drug absorption

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Bundang, Gyeonggi-do, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Period 1 : A (Amlodipine 10mg PO single dose) Period 2 : L (Losartan 100mg PO single dose) Period 3 : ALC (Amlodipine 10mg + Losartan 100mg + Chlorthalidone 25mg PO single dose) Period 4 : C (Chlorthalidone 25mg PO single dose)
- Sequence 2: Period 1 : L (Losartan 100mg PO single dose) Period 2 : C (Chlorthalidone 25mg PO single dose) Period 3 : A (Amlodipine 10mg PO single dose) Period 4 : ALC (Amlodipine 10mg + Losartan 100mg + Chlorthalidone 25mg PO single dose)
- Sequence 3: Period 1 : C (Chlorthalidone 25mg PO single dose) Period 2 : ALC (Amlodipine 10mg + Losartan 100mg + Chlorthalidone 25mg PO single dose) Period 3 : L (Losartan 100mg PO single dose) Period 4 : A (Amlodipine 10mg PO single dose)
- Sequence 4: Period 1 : ALC (Amlodipine 10mg + Losartan 100mg + Chlorthalidone 25mg PO single dose) Period 2 : A (Amlodipine 10mg PO single dose) Period 3 : C (Chlorthalidone 25mg PO single dose) Period 4 : L (Losartan 100mg PO single dose)
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 10 (A,C,ALC: intervention (8 days), L: intervention (4 days), Each period washout (14days)) | 7 (A,C,ALC: intervention (8 days), L: intervention (4 days), Each period washout (14days)) | 8 (A,C,ALC: intervention (8 days), L: intervention (4 days), Each period washout (14days)) | 8 (A,C,ALC: intervention (8 days), L: intervention (4 days), Each period washout (14days))
Completed | 7 | 7 | 6 | 6
Not Completed | 3 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: Period 1 : A Period 2 : L Period 3 : ALC Period 4 : C
- Sequence 2: Period 1 : L Period 2 : C Period 3 : A Period 4 : ALC
- Sequence 3: Period 1 : C Period 2 : ALC Period 3 : L Period 4 : A
- Sequence 4: Period 1 : ALC Period 2 : A Period 3 : C Period 4 : L
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Total
Number analyzed (Participants) | 10 | 7 | 8 | 8 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.70 (4.06) | 26.43 (4.89) | 26.00 (3.93) | 24.88 (4.05) | 26.06 (4.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 10 | 7 | 8 | 8 | 33
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 10 | 7 | 8 | 8 | 33

OUTCOME MEASURES:

1. Primary Outcome: AUClast
Description: AUClast(Area under the curve to the last measurable concentration)
Time Frame: 0, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 120, 168hr
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio(Comb/Alone)
Groups:
- HGP0904: HGP0904(amlodipine) ratio in single or combination
- HGP0608: HGP0608(losartan) ratio in single or combination
- HGP1405: HGP1405(chlorthalidone) ratio in single or combination
- EXP3174: EXP3174(losartan active metabolite) ratio in single or combination
Arm/Group | HGP0904 | HGP0608 | HGP1405 | EXP3174
Number analyzed (Participants) | 28 | 27 | 27 | 27
Ratio(Comb/Alone) | 1.0360 [0.9958 to 1.0778] | 1.1606 [1.0885 to 1.2375] | 1.0266 [0.9752 to 1.0807] | 1.0902 [1.0350 to 1.1148]

2. Primary Outcome: Cmax
Description: Cmax(maxium concentration)
Time Frame: 0, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 120, 168hr
Reporting Status: Not Posted

3. Secondary Outcome: AUCinf
Description: AUCinf(Area under the curve to infinity)
Time Frame: 0, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 120, 168hr
Reporting Status: Not Posted

4. Secondary Outcome: Tmax
Description: Tmax(Time to maximum concentration)
Time Frame: 0, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 120, 168hr
Reporting Status: Not Posted

5. Secondary Outcome: T1/2
Description: T1/2(Terminal elimination half-life),
Time Frame: 0, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 120, 168hr
Reporting Status: Not Posted

6. Secondary Outcome: CL/F
Description: CL/F(Apparent clearance)
Time Frame: 0, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 120, 168hr
Reporting Status: Not Posted

7. Secondary Outcome: Vz/F
Description: Vz/F(Apparent volume of distribution)
Time Frame: 0, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 120, 168hr
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Number of Paticipants With Adverse Events
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- HGP0904: amlodipine
  HGP0904
- HGP0608: losartan
  HGP0608
- HGP1405: chlorthalidone
  HGP1405
- HGP0904+HGP0608+HGP1405: amlodipine + losartan + chlorthalidone
  HGP0904
  HGP0608
  HGP1405
Arm/Group | HGP0904 | HGP0608 | HGP1405 | HGP0904+HGP0608+HGP1405
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/27 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/27 | 2/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HGP0904 (N=28) | HGP0608 (N=27) | HGP1405 (N=27) | HGP0904+HGP0608+HGP1405 (N=28)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HGP0904 (N=28) | HGP0608 (N=27) | HGP1405 (N=27) | HGP0904+HGP0608+HGP1405 (N=28)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No